CLINICAL TRIAL: NCT04731259
Title: A Phase 1b/2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety of ATR-04 to Reduce the Severity of Epidermal Growth Factor Inhibitor Associated Papulopustular Rash
Brief Title: Study to Evaluate the Safety of ATR-04
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons.
Sponsor: Azitra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTAR-403
Record Dates: First submitted 2021-01-14; First posted 2021-01-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Epidermal Growth Factor; Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATR-04 (Experimental): The intervention is an ointment that will be applied topically BID for 28 days. It will be supplied in small aluminum foil packets. Packets of study medication will be labeled with Subject Kit numbers to ensure the double-blind treatment.
  Interventions: Drug: ATR-04
- Placebo (Placebo Comparator): Placebo ointment will be applied topically BID for 28 days. It will be supplied in small aluminum foil packets. Packets of study medication will be labeled with Subject Kit numbers to ensure the double-blind treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ATR-04 — ATR-04 is a proprietary formulated product containing lyophilized SEΔΔΔ, a Staphylococcus epidermidis genetically modified to be auxotrophic to D-alanine as the active ingredient.
  Arms: ATR-04
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase 1b/2a study designed to evaluate the safety of an investigational product called ATR-04, to reduce the severity of epidermal growth factor receptor inhibitor (EGFRI) associated papulopustular rash on the face. This study will be performed at 10-12 clinical sites, with potentially a virtual component. Approximately 60 eligible subjects will participate. A subject's participation in the study will be up to a maximum of 86 days (up to 28 days for Screening, 28 days of BID treatment, and a 30 day no treatment follow-up period).

The primary objective of this study is to evaluate the safety and tolerability of ATR-04 compared to placebo.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled phase 1b/2a study designed to evaluate the safety of an investigational product called ATR-04 to reduce the severity of epidermal growth factor receptor inhibitor (EGFRI) associated papulopustular rash on the face. This study will be performed at 10-12 clinical sites, with potentially a virtual component. After informed consent is obtained, subjects will enter a screening period for up to 28 days to determine eligibility prior to randomization.

Approximately 60 eligible subjects, will be randomized to receive ATR-04 or a placebo, in a ratio of 1:1.

On Day 1, subjects will be instructed on study medication administration technique, the first application by the subject will be observed in person, via telehealth or via video connection and the subject will be monitored for adverse events (AEs) for at least 20 minutes.

Subjects will perform twice daily (BID) study assigned medication applications for 28 days. Subjects will have in person or virtual visits throughout the study. Subjects will return all study materials (i.e. diary cards, and study medication containers, swabs) either in person or via mail on Day 29 for their End of Treatment visit.

Beginning on Day 1, subjects will be assessed for safety. In addition, subjects' faces will be examined and assessed utilizing the Investigator Global Assessment (IGA) in person or via a virtual visit. Subjects will complete the Quality of Life (QoL) tool and standardized digital photographs will be taken.

A subject's participation in the study will be up to a maximum of 86 days (up to 28 days for Screening, 28 days of BID treatment, and a 30 day no treatment follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age inclusive, at the time of signing the informed consent
* Subjects with a current diagnosis of cancer
* IGA grade of 0 on the face
* Life expectancy, in the Investigator's opinion, greater than 12 weeks
* Plan to initiate treatment with one of the following EGFRI drugs (other treatments may be considered after consultation with the Sponsor): Cetuximab or Panitumumab or erlotinib
* Able to use Dove sensitive skin body wash for the duration of the treatment period.
* Acceptable and willing to delay start of EGFRI therapy until study eligibility is determined
* Anticipated to continue EGFRI therapy for at least 28 days after the first application of study medication
* Male and/or female
* Contraceptive use by men or women consistent with the EGFRI treatment package insert regarding the methods of contraception for those participating in clinical studies
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the study protocol.

Exclusion Criteria:

* Active bacterial skin infections on the face
* Inter-current illness that in the Investigator's opinion puts the subject at undue risk by study participation or interfere with the study conduct or evaluations
* Pregnant women
* EGFRI therapy within the previous 12 weeks
* Radiation therapy exposure to the face within the previous 8 weeks
* Use of topical steroids on the face within the previous 4 weeks
* Use of systemic antibiotics or topical antibiotics on the face in the previous 7 days
* Participation in an investigational clinical study in which administration of an investigational study medication occurred with the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), incidence of abnormal laboratory values, abnormal physical exams and abnormal vital signs. | Through study completion, on average of 1 year
  Safety and tolerability of ATR-04 compared to placebo as assessed by incidence and severity of Adverse Events (AEs), Serious Adverse Events (SAEs), laboratory values, physical exams and vital signs.

SECONDARY OUTCOMES:
Efficacy of ATR-04 assessed by IGA. | Up to Day 29
  Assess the efficacy of ATR-04 compared to placebo to mitigate the severity of EGFRI-associated skin effects as assessed by IGA.
Proportion of Subjects with Moderate or Severe Rash | Up to Day 29
  Difference in proportion of subjects with moderate or severe facial rash as assessed by IGA.
Difference in Subjects That Require Additional Therapies | Up to Day 29
  Difference in number of subjects that require additional therapies for the facial rash, such as antibiotics or steroids for ATR-04 compared to placebo.
Difference in Quality of Life (QoL) of Subjects | Up to Day 58.
  Difference in QoL of subjects on ATR-04 compared to placebo as assessed by FACT-EGFRI-18. Score ranges from 0-72, with higher scores indicating better outcomes.
Difference in Number of Inflammatory Lesions | Up to Day 29.
  Difference in number of inflammatory lesions on face for subjects on ATR-04 compared to placebo.
Difference in Proportion of Subjects That Stop/Decrease EGFRI Therapy | Up to Day 29.
  Difference in proportion of subjects that stop or decrease dose of EGFRI therapy.

OTHER OUTCOMES:
Exploratory Endpoint to Evaluate Change in EGFRI Skin Rash Microbiome | Through study completion, on average of 1 year
  Evaluate the microbiome of EGFRI skin rashes as determined by shotgun sequencing.
Exploratory Endpoint to Evaluate the Change in Skin Microbiome Associated with EGFRI Therapy | Through study completion, on average of 1 year
  Evaluate the change in skin microbiome associated with EGFRI therapy as determined by shotgun sequencing.

IPD SHARING:
Plan to Share IPD: No